CLINICAL TRIAL: NCT00570336
Title: A Dose Response Study of CTS-1027 in Hepatitis C Patients
Brief Title: Study of CTS-1027 in Hepatitis C Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Conatus Pharmaceuticals Inc. (Industry)
Collaborators: FGK Clinical Research GmbH (Industry)
Responsible Party: MiRa Huyghe, Conatus Pharmaceuticals Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTS-1027-01
Record Dates: First submitted 2007-12-06; First posted 2007-12-10 (Estimated); Last update posted 2010-09-16 (Estimated); Status verified 2010-09

CONDITIONS: Chronic Hepatitis C Virus Infection
Keywords: HCV; HCV treatment failure; Elevated aminotransferases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 2.5 milligram (mg) CTS-1027 (Experimental): 2.5 mg CTS-1027
  Interventions: Drug: CTS-1027
- 5 mg CTS-1027 (Experimental): 5 mg CTS-1027
  Interventions: Drug: CTS-1027
- 10 mg CTS-1027 (Experimental): 10 mg CTS-1027
  Interventions: Drug: CTS-1027
- 30 mg CTS-1027 (Experimental): 30 mg CTS-1027
  Interventions: Drug: CTS-1027
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CTS-1027 — Eligible patients were randomized to one of four doses of CTS-1027 (2.5 mg, 5 mg, 10 mg, or 30 mg) or placebo qd (quaque die, once daily).
  Arms: 10 mg CTS-1027; 2.5 milligram (mg) CTS-1027; 30 mg CTS-1027; 5 mg CTS-1027
Other: Placebo — Eligible patients were randomized to one of four doses of CTS-1027 (2.5 mg, 5 mg, 10 mg, or 30 mg) or placebo qd.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if CTS-1027 can lower elevated liver enzymes in patients with chronic HCV infection.

DETAILED DESCRIPTION:
Randomized, placebo-controlled, double-blind, parallel group, multicenter, dose response trial utilizing four doses of CTS-1027, administered orally once daily, in outpatients with chronic hepatitis C virus (HCV) infection.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients of minimum adult legal age (according to local laws for signing the informed consent document), able to provide written informed consent, and understand and comply with the requirements of the trial
* A history of chronic HCV infection
* Unsuccessful HCV treatment defined as one or more of the following criteria:

  1. Failure to achieve a virologic response during previous therapy, or
  2. Failure to tolerate therapy, or
  3. Failure to maintain a sustained virologic response, or
  4. In the opinion of the Principal Investigator, the patient is not a suitable candidate for interferon based therapy
* Liver impairment, as defined by either aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) levels 1.5 - 7 x ULN on at least two occasions, seven or more days apart, during the baseline period
* Alpha-fetoprotein (AFP) <= 50 ng/mL
* Hemoglobin >= 10 g/dL, platelet count >= 75 x 109/L, and white blood cell count >= 1.5 x 109/L
* Willingness to utilize adequate contraception (if female, evidenced by being postmenopausal for at least 6 months or using contraceptive pill; for both females and males, being surgically sterile, or using two forms of barrier contraception) from screening to at least one month after the completion of the trial.

Exclusion Criteria:

* Decompensated or severe liver disease defined by one or more of the following criteria:

  1. Prior liver biopsy showing cirrhosis
  2. Prior liver biopsy showing bridging fibrosis (Metavir >2 or Ishak >3) more than 2 years ago in the absence of newer liver biopsy results
  3. Prothrombin time: 3 seconds > control
  4. Total bilirubin >= 1.5 x Upper limit of the normal range (ULN), or > 3 x ULN for unconjugated bilirubin
  5. Serum albumin below normal limits
  6. AST or ALT > 7 x ULN during baseline period
  7. Evidence of portal hypertension including:
* Splenomegaly or evidence of portal hypertension (i.e., enlarged portal vein and varices) on ultrasound,
* Varices in esophagogastroduodenoscopy (EGD); or
* Ascites
* Hepatocellular carcinoma (HCC) or suspicion of HCC clinically or on ultrasound (or other imaging techniques)
* Known history or presence of human immunodeficiency virus (HIV) infection
* Co-infection with hepatitis B virus (HBV)
* If female: pregnant, lactating, or positive serum or urine pregnancy test
* Last baseline AST and ALT level prior to Day 1 of < 1.5 x ULN
* Renal impairment (creatinine > 1.5 x ULN) or hepatorenal syndrome
* Pancreatitis
* Hospitalization for liver disease within 60 days of screening
* Use of concomitant or prior drug therapy for HCV at screening, including the use of:

  1. drugs with presumed anti-HCV activity in the prior three months
  2. corticosteroids in the past 30 days
  3. potentially hepatotoxic drugs in the past 30 days (including alpha methyl-dopa, sodium valproic acid, isoniazide, or nitrofurantoin)
* Use of illicit or drugs of abuse in the prior three months (allowed if medically prescribed or indicated)
* History of alcohol abuse within the past year
* History or presence of clinically concerning cardiac arrhythmias or prolongation of pre-dose QT or QTc interval of > 450 milliseconds
* Other concomitant disease or condition likely to significantly decrease life expectancy (e.g., moderate to severe congestive heart failure) or any malignancy other than curatively treated skin cancer (basal cell or squamous cell carcinomas), unless adequately treated or in complete remission for ten or more years
* Any patient who has received any investigational drug or device within 30 days of dosing, or who is scheduled to receive another investigational drug or device during the course of this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2007-12; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Number of adverse events at each dose level | 4 to 24 weeks
Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) levels at each dose | 4-24 Weeks

SECONDARY OUTCOMES:
Peak and trough levels of CTS-1027 in plasma | 4 to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: William Frank, MD, Study Director — Conatus Pharmaceuticals Inc.
Locations (19):
- United States (19):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Scripps Clinic, La Jolla, California
  - Kaiser Permanente, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - University of Colorado Denver, Aurora, Colorado
  - University of Miami, Miami, Florida
  - Digestive Healthcare of Georgia, Atlanta, Georgia
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Health System, West Bloomfield, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Mt. Sinai School of Medicine, New York, New York
  - Bronx VA Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Consultants of Clinical Research, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Advanced Liver Therapies - Baylor College of Medicine, Houston, Texas
  - VAMC - Baylor College of Medicine, Houston, Texas
  - McGuire Hospital DVAMC, Richmond, Virginia